CLINICAL TRIAL: NCT00664742
Title: The Effect Of Fluvastatin XL® Treatment On The Lipid Profile In Patients With Metabolic Syndrome
Brief Title: The Effect of Fluvastatin XL® Treatment in Patients With Metabolic Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Medical Affairs, Novartis Pharmaceuticals
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CXUO320BTR03
Record Dates: First submitted 2008-04-21; First posted 2008-04-23 (Estimated); Results first posted 2011-05-17 (Estimated); Last update posted 2011-05-17 (Estimated); Status verified 2011-04

CONDITIONS: Metabolic Syndrome
Keywords: Metabolic syndrome,dyslipidemia,fluvastatin extended release
MeSH Terms: conditions — Metabolic Syndrome | interventions — Fluvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fluvastatin XL® Treatment (Experimental): 80 mg once daily, at bedtime.
  Interventions: Drug: Fluvastatin XL®

INTERVENTIONS:
Drug: Fluvastatin XL® — Fluvastatin extended release 80 mg
  Other Names: Lescol XL

SUMMARY:
This study evaluated safety, tolerability and efficacy of Fluvastatin XL® -extended release (80 mg once daily) in patients with metabolic syndrome

ELIGIBILITY:
Inclusion Criteria:

* ≥ 3 criteria for metabolic syndrome National Cholesterol Education Program Adult Treatment Panel III (NCEP ATP III criteria)
* Triglyceride (TG) < 400 mg/dl and Low Density Lipoprotein-Cholesterol (LDL-C) 100 mg/dl to 190 mg/dl
* Written informed consent for participating in the study

Exclusion Criteria:

* Severe renal disease or renal dysfunction
* Chronic liver disease or liver function impairment
* Inflammatory muscle dysfunction or findings of muscle problems
* Severe cardiac failure

Other protocol defined inclusion exclusion criteria may apply

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 614 (Actual)
Dates: Start 2006-09; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Götzepe Education and Research Hospital, Istanbul, Turkey (Türkiye)

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 614 participants enrolled. 607 participants treated.
Period: Overall Study
Arm/Group | Fluvastatin XL® Treatment
Started | 607
Completed | 481
Not Completed | 126
Not completed — Withdrawn due to adverse events | 3
Not completed — Withdrawal by Subject | 31
Not completed — Lost to Follow-up | 92

BASELINE CHARACTERISTICS:
Arm/Group | Fluvastatin XL® Treatment
Number analyzed (Participants) | 607
Age Continuous [Mean (Standard Deviation); unit: years] | 54 (10)
Sex/Gender, Customized [Number; unit: participants]
  Female | 421
  Male | 183
  Gender not recorded | 3

OUTCOME MEASURES:

1. Primary Outcome: Change in Total Cholesterol (TC), High Density Lipoprotein-Cholesterol (HDL-C), Low Density Lipoprotein-Cholesterol (LDL-C) and Triglycerides (TG) Levels From Baseline to Week-6
Description: Mean Absolute change in lipid profile parameters (TC, HDL-C, LDL-C and TG) calculated by the mean level for each parameter at week 6 minus the mean level at baseline.
Time Frame: Baseline,6 weeks
Population: The analysis was done on the Per Protocol Population which consists of all participants who did not violate inclusion/ exclusion criteria, completed the treatment study phase or withdrew from the study due to progression, death, or toxicity (AE related to study drug) and had at least one key response evaluation.
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Fluvastatin XL® Treatment
Number analyzed (Participants) | 481
mg/dL
  Change in TC | -50.4 (28.99897) [-53.4 to -47.5]
  Change in HDL-C | -0.6 (12.30119) [-1.4 to 0.2]
  Change in LDL-C | -45.2 (62.92132) [-47.7 to -42.8]
  Change in TG | -22.3 (71.50801) [-27.9 to -16.7]

2. Secondary Outcome: Percentage of Participants Achieving Total Cholesterol (TC), Low Density Lipoprotein-Cholesterol (LDL-C), High Density Lipoprotein-Cholesterol (HDL-C) and Triglycerides (TG) Predefined Target Lipid Levels
Description: The percentage of participants who achieved the following predefined lipid target levels at Baseline and at 6 months: TC <200 mg/dL, LDL-C <100 mg/dL, HDL-C >=60 mg/dL and TG < 150 mg/dL.
Time Frame: Baseline, 6 weeks
Population: This analysis was done on the safety population which consists of all participants who received at least one dose of study medication.
Measure: Number; unit: Percentage of Participants
Arm/Group | Fluvastatin XL® Treatment
Number analyzed (Participants) | 607
Percentage of Participants
  TC<200 mg/dL at Baseline | 22.4
  TC<200 mg/dL at Week-6 | 64.9
  LDL-C < 100 mg/dL at Baseline | 0.7
  LDL-C < 100 mg/dL at Week-6 | 51.2
  HDL-C >= 60 mg/dL at Baseline | 13.7
  HDL-C >= 60 mg/dL at Week-6 | 10.0
  TG < 150 mg/dL at Baseline | 33.6
  TG < 150 mg/dL at Week-6 | 39.5

ADVERSE EVENTS:
Time Frame: 6 Weeks
Arm/Group | Fluvastatin XL® Treatment
Serious Adverse Events (participants affected / at risk) | 2/607
Other Adverse Events (participants affected / at risk) | 0/607
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fluvastatin XL® Treatment (N=607)
Rhabdomyolysis and Myalgia (Musculoskeletal and connective tissue disorders) | 1
Coronary Artery Bypass Surgery (Cardiac disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.